CLINICAL TRIAL: NCT05296941
Title: Screening for Oral Cancer for Early Detection of Premalignant Disorders
Brief Title: Oral Cancer Screening for Early Detection of Premalignant Disorders (PMOD)
Acronym: PMOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna County Council, Sweden (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Kristina Edman, PhD, Dalarna County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Public dental care
Record Dates: First submitted 2022-03-08; First posted 2022-03-25 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Mouth Neoplasms
Keywords: oral cancer; potentially malignant disorders; leukoplakia; erythroplakia; oral lichen planus
MeSH Terms: conditions — Mouth Neoplasms; Leukoplakia; Erythroplasia; Lichen Planus, Oral

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brush biopsy (Experimental): Brusch biopsy at baseline and at 3 or 6 months
  Interventions: Procedure: Brush sampling
- Care as usual (Active Comparator): Control at 3 or 6 month, surgical biopsy when needed
  Interventions: Procedure: Brush sampling

INTERVENTIONS:
Procedure: Brush sampling — Brush sampling instead of surgical biopsy for control of reaccurance

SUMMARY:
Cancer is a complex disease; its different causes and types have a strong impact on patient treatment and prognosis. To improve understanding of the disease, its causes and progression, the investigators will develop a simple, cost-effective system for continuous control of mucosal lesions with non-invasive brush biopsy that can be managed in primary dental care, as an alternative to tissue biopsy in order to reduce the number of oral cavity cancers.

DETAILED DESCRIPTION:
In Sweden, about 1,200 cases of cancer of the oral cavity, lips and throat are diagnosed each year. This is significantly higher than the global age-standardized incidence of 6.1 per 100,000 inhabitants, including all ages and genders. Oral cancer is a serious and growing public health problem and leads to significantly reduced quality of life after extensive treatment that usually includes radiation therapy and surgery. Patients often have pain, swallowing problems, dry mouth that causes tooth status, negatively affected appearance, family life and social interaction. Although it is well known that early diagnostic screening is of great importance for increasing survival, there is a lack of a nationally organized screening program of high-risk individuals, tobacco users and individuals with overconsumption of alcohol. As a result, many cases are diagnosed late and therefore have poor prognosis. The five-year survival rate in Sweden for the diagnosis of oral cancer is about 60%. If the tumor is small when diagnosed, without lymph node involvement or metastases,and treated correctly, a survival rate of 90% can be achieved while in a late diagnosis with the presence of lymph node involvement and metastases, survival drops drastically and is only 36%. A large proportion of oral cancer originates from potentially malignant oral mucosal lesions (PMOD) that occur in a prevalence of about 2-3% globally and over time are at risk of malignification. Of PMOD, oral leukoplakia (OL) is the most prevalent and most common in the group of middle-aged or older men. Swedish prevalence figures for OL have been reported to range from 0.7% to 3.5%. As patients with PMOD such as OL, erythroplakia (EP) or proliferative verrukös are at a significantly increased risk of developing oral cancer, it is important to include these patients in a functioning control system. This is especially true for risk individuals, those with an overconsumption of alcohol, with tobacco use, and those with chronic infection of tonsil and tongue base with high-risk human papillomavirus. About 80% of the adult population in Sweden is regularly examined at private dental care or public dental care, which means that general dental care can take a great responsibility for identifying and carrying out continuous checks on risk groups. A routine examination of the patient should include assessment of the oral mucosa according to clinical practice. Oral mucosal changes should be diagnosed and, if necessary, treatment initiated. In the case of a clinical diagnosis of OL, EP or verrukös leukoplakia, the clinical diagnosis should be verified with a tissue biopsy performed at a specialist clinic in orofacial medicine, oral surgery or ear-nose-throat clinic. Based on the diagnosis and degree of cell changes, it is decided according to current practice whether the continued treatment and the patient is included in a system for continuous checks. Oral cancer must be diagnosed early because mortality is high, especially in late diagnosis, and quality of life after treatment is very poor with significant pain, speech, chewing and swallowing difficulties with a strong impact on both family life and social contacts and working life. The solution is early detection and early treatment, which can be achieved if follow-up are performed in primary dental care with non-invasive brush biopsies for cytological diagnostics in a similar way to cervical cancer screening managed by midwives. Cytological diagnosis of oral mucosal changes is a safe, simple and rapid method with high sensitivity and specificity. With the present series of studies, the investigators intend to evaluate different possibilities to identify PMOD with high-grade dysplasias, and tumors early in order to improve prognosis.

ELIGIBILITY:
Inclusion Criteria:

• Persons 18 years of age or older who have the clinical diagnosis of leukoplakia, erythroplakia or proliferative verrukös leukoplakia

Exclusion Criteria:

* People who cannot read and understand information in Swedish.
* Ongoing chemotherapy and/or radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Numbers of cancers diagnosed by brush sampling | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Public dental care, Principal Investigator — Uppsala University
Locations (1):
- Kristina Edman, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided